CLINICAL TRIAL: NCT02014545
Title: Phase II Trial Evaluating the Addition of Lucanthone to Whole Brain Radiation Therapy in Patients With Brain Metastases From Non-Small Cell Lung Cancer
Brief Title: Evaluation of Lucanthone to Whole Brain Radiation Therapy in Patients With Brain Metastases From Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Pending resolution of study drug issues
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00037529; IRB00037529 (Other: CCCWFU)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Brain Metastases; Non-small Cell Lung Cancer
Keywords: brain metastases; non-small cell lung cancer; whole brain radiation therapy; lucanthone
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Lucanthone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WBRT + Lucanthone (Active Comparator): Treatment will consist of WBRT given in a dose of 30 Gy in ten fractions with lucanthone given as an adjunct. Lucanthone will be administered as 25 mg and 100 mg tablets to be swallowed. Dosage will be one of the following: 250 mg bid, 250 tid, or 375 mg tid.
  Interventions: Drug: Lucanthone
- WBRT + Placebo (Placebo Comparator): Patients will receive prophylactic cranial irradiation at 3 Gy per fraction, 5 days per week, for 2 weeks to a total dose of 30 Gy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lucanthone — The dose of lucanthone to be administered will be calculated based on the patient's body weight. The dose to be given will be 250 bid, 250 tid or 375 tid dependent upon study progression.
  Arms: WBRT + Lucanthone
Other: Placebo — Only standard treatment of whole brain radiation therapy is done.
  Arms: WBRT + Placebo

SUMMARY:
This is a randomized, double blind placebo controlled study to evaluate safety and efficacy of lucanthone administered as an adjunct to patients receiving whole brain radiation therapy (WBRT) as primary treatment for brain metastases secondary to non-small cell lung cancer.

DETAILED DESCRIPTION:
Eligible patients for this trial will be randomized to lucanthone or placebo in a ratio of 1:1. The treatment will consist of WBRT given in a dose of 30 Gy in ten fractions. Lucanthone/placebo will be given as an adjunct to the WBRT on days that WBRT is administered. Tumor assessments will be done with a brain MRI. Radiological assessments on the tumor will be made periodically throughout the study and will be discontinued at the time of tumor progression. Safety will be evaluated for one year during the study period and survival data will be collected thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given informed consent.
* The patient is willing and able to abide by the protocol.
* The patient is between age 18 and 70 (between 19 and 70 in Alabama).
* The patient has histologically proven NSCLC with radiologically documented brain metastases.
* Newly diagnosed or stable systemic disease, on or off systemic therapy.
* If receiving systemic therapy for NSCLC, at least two weeks since patient received systemic therapy.
* Able to withhold systemic therapy for duration of WBRT therapy.
* If the patient is of childbearing potential, he/she is using an acceptable/effective method of contraception.
* The patient's Karnofsky Score is greater than or equal to 70%.

Exclusion Criteria:

* Patient has a diagnosis of recurrent brain metastases.
* The patient has an absolute neutrophil count less than or equal to 1.5 X 10 9/L.
* The patient has a screening platelet count less than 100,000/uL.
* The patient has a screening bilirubin greater than 1.6 mg/dL.
* The patient has a screening creatinine greater than 2.25 mg/dL in men and 1.8 mg/dL in women.
* The patient has a screening ALT/AST greater than 2.5 times the upper limit of the laboratory reference range.
* The patient has an unstable medical condition or significant comorbid pathophysiology (e.g. active infection, poorly controlled diabetes, unstable angina, severe heart failure) that would interfere with his/her participation in the study.
* The patient is enrolled, or plans to enroll, in a concurrent treatment protocol with another investigational product.
* The patient has received prior chemotherapy or radiation therapy within two weeks of beginning WBRT on protocol.
* The patient is allergic to gadolinium contrast.
* More than 21 days has or will elapse between the brain MRI documenting the brain metastases and the initiation of WBRT.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of lucanthone when given during WBRT | 2 weeks to 13 months
  Progression free survival at 6 months and one year, overall response rate at months 1, 4, 7, 10, and 13 months and overall survival at 13 months will be evaluated. MRI brain scans will be performed baseline and months 1, 4, 7, 10, and 13. Objective assessments of overall response will be based on tumor assessments from MRI scans interpreted using the Revised Assessment in Neuro-Oncology (RANO) criteria.

SECONDARY OUTCOMES:
Evaluate the safety and toxicity of lucanthone when used in combination with standard doses of WBRT in the primary treatment of brain metastases secondary to non-small cell lung cancer | 2 weeks to 13 months
  Safety will be monitored throughout the study by physical exams, review of adverse events, and laboratory studies.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan C. Grant, MD, JD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States